CLINICAL TRIAL: NCT04676802
Title: Pain Relief After Trapeziectomy Without Opioids: Ibuprofen & Acetaminophen Versus Oxycodone
Brief Title: Pain Relief After Trapeziectomy: Ibuprofen & Acetaminophen Versus Oxycodone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amy Ladd, Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 58972
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pain, Postoperative; Osteoarthritis Thumb
MeSH Terms: conditions — Pain, Postoperative | interventions — Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSAIDS (Experimental): Following surgery will receive NSAID capsules following surgery. Will take online and phone surveys.
  Interventions: Drug: NSAID capsules
- Opioids (Experimental): Following surgery will receive opioid capsules following surgery. Will take online and phone surveys.
  Interventions: Drug: Opioid capsule

INTERVENTIONS:
Drug: NSAID capsules — 1, Ibuprofen 400-mg and 1, Acetaminophen 500-mg capsule per dosage
  Arms: NSAIDS
Drug: Opioid capsule — 1, Oxycodone 5-mg capsule and 1, placebo capsule per dosage
  Arms: Opioids

SUMMARY:
In the US, pain management after surgery for surgical treatment of osteoarthritis at the base of the thumb typically consists of prescription opioids during the early recovery phase. Given the highly addictive nature of prescription opioids, guidelines are being evaluated by hand surgeons to reduce opioid use while still maintaining pain control after surgery. A promising approach is to use non-narcotic medication as the first line of treatment. The purpose of this study is to demonstrate the efficacy of a combination of non-steroidal anti-inflammatory drugs (NSAIDs), ibuprofen and acetaminophen, in comparison to a morphine analogue substance (oxycodone) for pain management in the first 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing trapeziectomy for thumb osteoarthritis

English proficient,

Exclusion Criteria:

* Pregnancy

Current use of opioids

Concurrent surgeries (ex. trapeziectomy combined with carpal tunnel release)

Inability to complete study forms (education, cognitive ability, mental status, medical status)

Allergy or intolerance to Ibuprofen, Acetaminophen and/or Oxycodone

Liver or kidney dysfunction, abnormal liver enzymes restricting use of acetaminophen or ibuprofen

History of chronic heart failure, upper gastrointestinal bleeding or coagulopathy

History of complex regional pain syndrome

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2021-12-27 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change of medication consumption and overall amount | Every day from the first day after surgery to 30 days post-op.
  The number of capsules consumed in the last 24 hours. Consumption rate and overall consumption will be compared between groups to assess efficacy and inform further statistical analyses.
Change of worst daily pain score measured over time | Every day from the first day after surgery to 30 days post-op.
  Numerical score describing surgical pain at its worst in the last 24 hours, between 1 and 10, 1 being no pain, 10 being the worst possible pain.
Change of least daily pain score measured over time | Every day from the first day after surgery to 30 days post-op.
  Numerical score describing surgical pain at its least in the last 24 hours, between 1 and 10, 1 being no pain, 10 being the worst possible pain.
Change of average daily pain score measured over time | Every day from the first day after surgery to 30 days post-op.
  Numerical score describing average surgical pain in the last 24 hours, between 1 and 10, 1 being no pain, 10 being the worst possible pain.

SECONDARY OUTCOMES:
Change in Quick DASH scores over time | Baseline, Post-operative weeks 1, 3, 5, and 8
  Quick Disabilities of the Arm, Shoulder, and Hand (qDASH) is a responsive measure to patient-reported functional change in the hand and upper extremity patient population, ranging from 0 to 100. Lower scores signify limited function and increased pain.
Change in PROMIS-PI scores over time | Baseline, Post-operative weeks 1, 3, 5, and 8
  PROMIS-PI scores (Patient-Reported Outcomes Measurement Information System - Pain Interference) are effective measures of the change in perceived pain, supporting intervention related studies assessing power analyses for comparative research.
  We use the Pain Interference - Short Form version 6b, which consists of 6 questions regarding how much the pain experienced in the last 7 days interfered with everyday aspects of life (i.e. enjoyment, ability to concentrate, day to day activities, recreational activities, doing tasks away from home, and socializing with others). The answers to all questions are ordinals ranging from 1 (not interfered at all) to 5 (interfered very much).

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ladd, MD, Principal Investigator — Stanford Orthopaedic Surgery
Locations (2):
- United States (2):
  - Stanford Health Care, Redwood City, California
  - University of Utah Health Care, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No